CLINICAL TRIAL: NCT05605834
Title: Assessment of Peroxide Level in Saliva During Teeth Bleaching With 9.5% Hydrogen Peroxide Gel Using a Tray With Reservoir Versus a Tray Without Reservoir. A Randomized Clinical Trial
Brief Title: Assessment of Peroxide Level in Saliva During Teeth Bleaching With 9.5% Hydrogen Peroxide Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Anas Yousef Mohammad, bachelor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: a tray with reservoir
Record Dates: First submitted 2022-10-29; First posted 2022-11-04 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Consumption; Toxicity
Keywords: hydrogen peroxide; reservoir; peroxide level; saliva; assessment; non reservoir

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen peroxide 9.5% bleaching using a tray with reservoir. (Experimental): 9.5% hydrogen peroxide bleaching (POLA DAY advanced tooth whitening system, SDI) using a tray with reservoir.
  Interventions: Other: 9.5% hydrogen peroxide bleaching (POLA DAY advanced tooth whitening system, SDI) using a tray with reservoir
- Hydrogen peroxide 9.5% bleaching using a tray without reservoir. (Active Comparator): 9.5% hydrogen peroxide bleaching (POLA DAY advanced tooth whitening system, SDI) using a tray without reservoir.
  Interventions: Other: 9.5% hydrogen peroxide bleaching (POLA DAY advanced tooth whitening system, SDI) using a tray without reservoir.

INTERVENTIONS:
Other: 9.5% hydrogen peroxide bleaching (POLA DAY advanced tooth whitening system, SDI) using a tray with reservoir — Patients will be randomly divided into two groups. Alginate impressions of maxillary dental arches of patients will be taken to obtain casts and produce the customized trays.
  Reservoirs 1 mm thick will be created on the facial surfaces of anterior teeth, including the first premolars in the arches, applying a light-cured resin on the casts. The resin layer thickness will be standardized using a thickness gauge (1.5 mm thickness). Then, customized trays will be fabricated with 0.9-mm-thick vinyl acetate sheets using the thermoforming process. Trays will be precisely trimmed completely involving tooth surface (1 mm incisal or occlusal to gingival margin), and the adaptation will be verified on the casts. The trays will be placed over teeth to verify the adaptation in the patients' mouth.
  Arms: Hydrogen peroxide 9.5% bleaching using a tray with reservoir.
Other: 9.5% hydrogen peroxide bleaching (POLA DAY advanced tooth whitening system, SDI) using a tray without reservoir. — Alginate impressions of maxillary dental arches of patients will be taken to obtain casts to produce the customized trays. Then, customized trays will be fabricated with no space for reservoir, with 0.9-mm-thick vinyl acetate sheets using the thermoforming process applying a light-cured resin on the casts. Trays will be precisely trimmed completely involving tooth surface (1 mm incisal or occlusal to gingival margin), and the adaptation will be verified on the casts. The trays will be placed over teeth to verify the adaptation in the participants' mouths.
  Arms: Hydrogen peroxide 9.5% bleaching using a tray without reservoir.

SUMMARY:
Assessment of peroxide level in saliva during teeth bleaching with 9.5% hydrogen peroxide gel using a tray with reservoir versus a tray without reservoir. A randomized clinical trial

DETAILED DESCRIPTION:
Statement of the Problem

There is more concern about the possible adverse effect of bleaching agent, patients report gastrointestinal mucosal irritation e.g. a burning palate, throat and minor upsets in the stomach and intestine. Some adverse effects of hydrogen peroxide as a dental bleaching agent include dentin sensitivity and/or gingival irritation led by unstable and reactive H+ free radicals and low pH from prolonged use. Peroxide is a highly reactive substance which can damage oral soft tissues and hard tissues when present in high concentrations and with exposures of prolonged duration. Several researches have focused on the problem of gel ingestion and potential peroxide release in saliva

Rationale

Reservoirs are modifications in the tray molds to increase the amount of bleaching material carried by the bleaching tray, seeking greater bleaching efficacy. The use of reservoirs in the bleaching trays was initially seen as positive, since higher accumulation of material could provide the patient with greater treatment efficacy. stated that there is no significant difference between groups whitened with and without reservoirs for gingival irritation or tooth sensitivity. Most authors and bleaching gel manufacturers recommend the use of reservoirs to increase the amount of product available for bleaching and to allow for complete seating of the bleaching tray, although that the reservoirs decrease tray retention and increase lab fabrication time and cost. The presence of reservoirs decreases the retention of the tray, allowing more room for the gel but also reducing the adaptation of the tray. That may cause more leakage of the material, which may lead to more peroxide level in saliva. A major concern for clinicians was the potential toxicological effect of hydrogen peroxide contacting soft tissues. A safe hydrogen peroxide exposure level (no observed effect level) was determined with catalase-deficient mice, reporting a maximum dose of 26 mg/kg/d. This corresponds to the dose level in humans, considering the conventional uncertainty factor of 100-fold, of 0.26 mg/kg/d . The safety of hydrogen peroxide products used for at home bleaching regarding peroxide release in saliva has not been fully proven.

ELIGIBILITY:
Inclusion Criteria:

* participants:

  1. Good general health.
  2. Adult patients aged 18-40 years.
  3. Absence of non-carious cervical lesions, active caries, gingival recession, or periodontal disease.
  4. Do not use orthodontics appliance or removable prosthesis.

teeth:

1. Maxillary anterior teeth without caries, restorations and/or endodontic treatment.
2. Mild generalized staining.

Exclusion Criteria:

* participants:

  1. Smoking or alcohol dependent patients.
  2. Pregnancy and lactating women.
  3. Parafunctional habits or pathologies.
  4. Periapical alterations.
  5. Use of medicaments that alter salivary flow.
  6. Patients who had already undergone tooth bleaching
  7. Patients with severe internal tooth discoloration as tetracycline stain, fluorosis or endodontic treatment.

teeth:

1. Tooth hypersensitivity.
2. Presence of cracks or fractures.
3. Periodontal affection sign and symptoms.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Peroxide level in saliva | T0: 1 min after beginning of the bleaching procedure and application of the tray
  Peroxide concentration in saliva (mg/ml)
Peroxide level in saliva | T1: 5 min after tray application
  Peroxide concentration in saliva (mg/ml)
Peroxide level in saliva | T2: 10 min after tray application
  Peroxide concentration in saliva (mg/ml)
Peroxide level in saliva | T3: 30 min after tray application
  Peroxide concentration in saliva (mg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Iman Ibrahim El Sayad, prof, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, Cairo, Egypt

REFERENCES:
- [Background] Alqahtani MQ. Tooth-bleaching procedures and their controversial effects: A literature review. Saudi Dent J. 2014 Apr;26(2):33-46. doi: 10.1016/j.sdentj.2014.02.002. Epub 2014 Mar 12. PMID 25408594
- [Background] Auschill TM, Hellwig E, Schmidale S, Sculean A, Arweiler NB. Efficacy, side-effects and patients' acceptance of different bleaching techniques (OTC, in-office, at-home). Oper Dent. 2005 Mar-Apr;30(2):156-63. PMID 15853099
- [Background] Bernardon JK, Sartori N, Ballarin A, Perdigao J, Lopes GC, Baratieri LN. Clinical performance of vital bleaching techniques. Oper Dent. 2010 Jan-Feb;35(1):3-10. doi: 10.2341/09-008CR. PMID 20166405
- [Background] Dahl JE, Pallesen U. Tooth bleaching--a critical review of the biological aspects. Crit Rev Oral Biol Med. 2003;14(4):292-304. doi: 10.1177/154411130301400406. PMID 12907697
- [Background] Marques DN, da Mata AD, Silveira JM, Marques JR, Amaral JP, Guilherme NF. Hydrogen peroxide release kinetics into saliva from different whitening products: a double-blind, randomized clinical trial. Clin Oral Investig. 2012 Feb;16(1):155-63. doi: 10.1007/s00784-010-0491-x. Epub 2011 Jan 8. PMID 21221681
- [Background] Geisinger S, Kwon SR, Qian F. Employment of Reservoirs in At-Home Whitening Trays: Efficacy and Efficiency in Tooth Whitening. J Contemp Dent Pract. 2015 May 1;16(5):383-8. doi: 10.5005/jp-journals-10024-1694. PMID 26162258
- [Background] Goldberg M, Grootveld M, Lynch E. Undesirable and adverse effects of tooth-whitening products: a review. Clin Oral Investig. 2010 Feb;14(1):1-10. doi: 10.1007/s00784-009-0302-4. Epub 2009 Jun 20. PMID 19543926
- [Background] Hannig C, Zech R, Henze E, Dorr-Tolui R, Attin T. Determination of peroxides in saliva--kinetics of peroxide release into saliva during home-bleaching with Whitestrips and Vivastyle. Arch Oral Biol. 2003 Aug;48(8):559-66. doi: 10.1016/s0003-9969(03)00102-x. PMID 12828984
- [Background] Hannig C, Zech R, Henze E, Dreier S, Attin T. Peroxide release into saliva from five different home bleaching systems in vivo. Am J Dent. 2005 Feb;18(1):13-8. PMID 15810475
- [Background] Hannig C, Willenbucher S, Becker K, Mahony C, Attin T. Recovery of peroxides in saliva during home bleaching--influence of smoking. J Oral Rehabil. 2006 Jul;33(7):533-41. doi: 10.1111/j.1365-2842.2005.01579.x. PMID 16774513
- [Background] Haywood VB. History, safety, and effectiveness of current bleaching techniques and applications of the nightguard vital bleaching technique. Quintessence Int. 1992 Jul;23(7):471-88. PMID 1410249
- [Background] Haywood VB, Leonard RH, Nelson CF, Brunson WD. Effectiveness, side effects and long-term status of nightguard vital bleaching. J Am Dent Assoc. 1994 Sep;125(9):1219-26. doi: 10.14219/jada.archive.1994.0154. PMID 7930184
- [Background] Haywood VB, Sword RJ. Tray bleaching status and insights. J Esthet Restor Dent. 2021 Jan;33(1):27-38. doi: 10.1111/jerd.12688. Epub 2020 Dec 5. PMID 33277968
- [Background] Javaheri DS, Janis JN. The efficacy of reservoirs in bleaching trays. Oper Dent. 2000 May-Jun;25(3):149-51. PMID 11203808
- [Background] Joiner A. The bleaching of teeth: a review of the literature. J Dent. 2006 Aug;34(7):412-9. doi: 10.1016/j.jdent.2006.02.002. Epub 2006 Mar 29. PMID 16569473
- [Background] Kirsten GA, Freire A, de Lima AA, Ignacio SA, Souza EM. Effect of reservoirs on gingival inflammation after home dental bleaching. Quintessence Int. 2009 Mar;40(3):195-202. PMID 19417883
- [Background] Kose C, Calixto AL, Bauer JR, Reis A, Loguercio AD. Comparison of the Effects of In-office Bleaching Times on Whitening and Tooth Sensitivity: A Single Blind, Randomized Clinical Trial. Oper Dent. 2016 Mar-Apr;41(2):138-45. doi: 10.2341/15-085-C. Epub 2015 Oct 28. PMID 26509229
- [Background] Li Y. Safety controversies in tooth bleaching. Dent Clin North Am. 2011 Apr;55(2):255-63, viii. doi: 10.1016/j.cden.2011.01.003. PMID 21473992
- [Background] Mailart MC, Sakassegawa PA, Torres C, Palo RM, Borges AB. Assessment of Peroxide in Saliva During and After At-home Bleaching With 10% Carbamide and Hydrogen Peroxide Gels: A Clinical Crossover Trial. Oper Dent. 2020 Jul 1;45(4):368-376. doi: 10.2341/19-127-C. PMID 32216723
- [Background] Martini EC, Favoreto MW, Coppla FM, Loguercio AD, Reis A. Evaluation of reservoirs in bleaching trays for at-home bleaching: a split-mouth single-blind randomized controlled equivalence trial. J Appl Oral Sci. 2020;28:e20200332. doi: 10.1590/1678-7757-2020-0332. Epub 2020 Aug 17. PMID 32813842
- [Background] Martini EC, Favoreto MW, de Andrade HF, Coppla FM, Loguercio AD, Reis A. One-year follow-up evaluation of reservoirs in bleaching trays for at-home bleaching. J Esthet Restor Dent. 2021 Oct;33(7):992-998. doi: 10.1111/jerd.12797. Epub 2021 Jul 1. PMID 34212493
- [Background] Matis BA, Hamdan YS, Cochran MA, Eckert GJ. A clinical evaluation of a bleaching agent used with and without reservoirs. Oper Dent. 2002 Jan-Feb;27(1):5-11. PMID 11817468
- [Background] Matis BA, Yousef M, Cochran MA, Eckert GJ. Degradation of bleaching gels in vivo as a function of tray design and carbamide peroxide concentration. Oper Dent. 2002 Jan-Feb;27(1):12-8. PMID 11817465
- [Background] Sulieman MA. An overview of tooth-bleaching techniques: chemistry, safety and efficacy. Periodontol 2000. 2008;48:148-69. doi: 10.1111/j.1600-0757.2008.00258.x. No abstract available. PMID 18715362
- [Background] Watt BE, Proudfoot AT, Vale JA. Hydrogen peroxide poisoning. Toxicol Rev. 2004;23(1):51-7. doi: 10.2165/00139709-200423010-00006. PMID 15298493
- [Background] Weiner ML, Freeman C, Trochimowicz H, de Gerlache J, Jacobi S, Malinverno G, Mayr W, Regnier JF. 13-week drinking water toxicity study of hydrogen peroxide with 6-week recovery period in catalase-deficient mice. Food Chem Toxicol. 2000 Jul;38(7):607-15. doi: 10.1016/s0278-6915(00)00048-x. PMID 10942322